CLINICAL TRIAL: NCT05606068
Title: A Novel Limb Cryocompression System for Prevention of Chemotherapy Induced Peripheral Neuropathy - Expansion Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Paxman Coolers Ltd. (Unknown); The N.1 Institute for Health, National University of Singapore (Unknown); Curie Oncology, Mount Elizabeth Novena Specialist Centre (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022/00486
Record Dates: First submitted 2022-10-25; First posted 2022-11-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Chemotherapy-induced Peripheral Neuropathy; Cryocompression

STUDY DESIGN:
Intervention Model Description: Cryocompression will be applied during every cycle of chemotherapy for a duration of up to 4 hours. All chemotherapy patients will receive 30 minutes pre-infusion cooling and 30 minutes post-infusion cooling. Cryocompression for each cycle will not exceed 4 hours. Chemotherapy and concomitant limb cryocompression are performed for 12 cycles and may be continued further in consultation with the PI. Overall, hypothermia will be administered for no longer than four hours.
  Each patient will undergo maximum limb cooling. The initial device settings for the first cycle for each patient will be based on the optimal temperature determined to be safe and tolerable in previous studies. The temperature will be adjusted according to the patient's tolerance/intolerance feedback during each cycle of cooling and documented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer patients (Experimental): Cancer patients will undergo limb cryocompression based on the established optimal temperature and pressure from previous studies over multiple cycles of chemotherapy to establish safety and tolerability of repeated therapy.
  Interventions: Device: Paxman Limb Cryocompression System (PLCS)

INTERVENTIONS:
Device: Paxman Limb Cryocompression System (PLCS) — The study population will comprise of cancer patients scheduled to receive weekly paclitaxel chemotherapy for a maximum of 12 cycles.
  Cryocompression will be applied during every cycle of chemotherapy for a duration of up to 4 hours. All chemotherapy patients will receive 30 minutes pre-infusion cooling and 30 minutes post-infusion cooling. Cryocompression for each cycle will not exceed 4 hours. Chemotherapy and concomitant limb cryocompression are performed for 12 cycles and may be continued further in consultation with the PI. Overall, limb cryocompression will be administered for no longer than four hours.

SUMMARY:
The study conducted on cancer patients is designed to test safety and efficacy of limb hypothermia in cancer patients using the new Paxman Limb Cryocompression System (PLCS). Ultimately this will lead to the development of a therapy regime that will help to prevent chemotherapy-induced neuropathy in cancer patients.

DETAILED DESCRIPTION:
The study will consist of 80 cancer patients, recruited from the National University Hospital and Curie Oncology. Based on an established optimal temperature and pressure of limb cryocompression, cancer patients will undergo cryocompression over multiple cycles of chemotherapy to establish safety and efficacy of repeated therapy. Cryocompression of the limbs will be administered using cooling wraps attached to a cooling device. The limbs will be cooled from the digits to the elbow/knee.

ELIGIBILITY:
Inclusion Criteria:

* Age 21- 80 years.
* Signed informed consent from patient or legal representative
* Scheduled to receive weekly paclitaxel chemotherapy
* Patients may receive other chemotherapy drugs alongside taxane e.g. Platinum/Herceptin.

Exclusion Criteria:

* Open skin wound or ulcers of the limbs
* History of Raynaud's phenomenon, peripheral vascular disease, or poorly controlled diabetes
* Pregnant woman
* A score of more than 5 in Total Neuropathy Score (TNS) at baseline for cancer patients

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events in cancer patients, over the duration of a limb cryocompression cycle, as assessed by Common Terminology Criteria for Adverse Events 5.0 | 4 months
  Defined as the number of patients with treatment-related intolerance as assessed by CTCAE v5.0. Grade 1-5 refer to the severity of the adverse event with higher grade indicating greater severity. Grade 3 and above will be considered severe.
Difference in qualitative symptom scores using the European Organisation of Research and Treatment of Cancer Quality of Life Questionnaire-CIPN twenty-item scale | 16 months
  Difference in qualitative symptom scores using the EORTC QLQ-CIPN-20 scale before, at the end of paclitaxel chemotherapy with limb cryocompression, and at 3,6 and 12 months post-treatment.
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy Module (EORTC QLQ-CIPN20) has 20 questions/items. This scale has a minimum of 1 and maximum of 4 for each of the 20 questions, with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
PLCS usability questionnaire | 4 months
  PLCS usability questionnaire will be given to patients after completing all 12 cycles of chemotherapy with cryocompression, to determine the tolerance level and user experience. The PLCS usability questionnaire has a total of 8 questions, some of which use a scale of 1 to 5, while other questions use a scale of 1 to 10. Some questions differ with regard to whether higher scores mean a better or worse outcome, but majority of the questions have higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Si Jing, Joline Lim, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - Curie Oncology, Mount Elizabeth Novena Specialist Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Windebank AJ, Grisold W. Chemotherapy-induced neuropathy. J Peripher Nerv Syst. 2008 Mar;13(1):27-46. doi: 10.1111/j.1529-8027.2008.00156.x. PMID 18346229
- [Background] Bandla A, Sundar R, Liao LD, Sze Hui Tan S, Lee SC, Thakor NV, Wilder-Smith EP. Hypothermia for preventing chemotherapy-induced neuropathy - a pilot study on safety and tolerability in healthy controls. Acta Oncol. 2016;55(4):430-6. doi: 10.3109/0284186X.2015.1075664. Epub 2015 Sep 11. PMID 26360921
- [Background] Sundar R, Bandla A, Tan SS, Liao LD, Kumarakulasinghe NB, Jeyasekharan AD, Ow SG, Ho J, Tan DS, Lim JS, Vijayan J, Therimadasamy AK, Hairom Z, Ang E, Ang S, Thakor NV, Lee SC, Wilder-Smith EP. Limb Hypothermia for Preventing Paclitaxel-Induced Peripheral Neuropathy in Breast Cancer Patients: A Pilot Study. Front Oncol. 2017 Jan 10;6:274. doi: 10.3389/fonc.2016.00274. eCollection 2016. PMID 28119855
- [Background] Bandla A, Tan S, Kumarakulasinghe NB, Huang Y, Ang S, Magarajah G, Hairom Z, Lim JSJ, Wong A, Chan G, Ngoi N, Ang E, Lee YM, Chan A, Lee SC, Thakor N, Wilder-Smith E, Sundar R. Safety and tolerability of cryocompression as a method of enhanced limb hypothermia to reduce taxane-induced peripheral neuropathy. Support Care Cancer. 2020 Aug;28(8):3691-3699. doi: 10.1007/s00520-019-05177-2. Epub 2019 Dec 6. PMID 31811482
- [Background] Loprinzi CL, Lacchetti C, Bleeker J, Cavaletti G, Chauhan C, Hertz DL, Kelley MR, Lavino A, Lustberg MB, Paice JA, Schneider BP, Lavoie Smith EM, Smith ML, Smith TJ, Wagner-Johnston N, Hershman DL. Prevention and Management of Chemotherapy-Induced Peripheral Neuropathy in Survivors of Adult Cancers: ASCO Guideline Update. J Clin Oncol. 2020 Oct 1;38(28):3325-3348. doi: 10.1200/JCO.20.01399. Epub 2020 Jul 14. PMID 32663120
- [Background] Jordan B, Margulies A, Cardoso F, Cavaletti G, Haugnes HS, Jahn P, Le Rhun E, Preusser M, Scotte F, Taphoorn MJB, Jordan K; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org; EONS Education Working Group. Electronic address: eons.secretariat@cancernurse.eu; EANO Guideline Committee. Electronic address: office@eano.eu. Systemic anticancer therapy-induced peripheral and central neurotoxicity: ESMO-EONS-EANO Clinical Practice Guidelines for diagnosis, prevention, treatment and follow-up. Ann Oncol. 2020 Oct;31(10):1306-1319. doi: 10.1016/j.annonc.2020.07.003. Epub 2020 Jul 30. No abstract available. PMID 32739407
- [Background] Stubblefield MD, Burstein HJ, Burton AW, Custodio CM, Deng GE, Ho M, Junck L, Morris GS, Paice JA, Tummala S, Von Roenn JH. NCCN task force report: management of neuropathy in cancer. J Natl Compr Canc Netw. 2009 Sep;7 Suppl 5:S1-S26; quiz S27-8. doi: 10.6004/jnccn.2009.0078. PMID 19755042
- [Background] Yeo F, Ng CC, Loh KWJ, Molassiotis A, Cheng HL, Au JSK, Leung KT, Li YC, Wong KH, Suen L, Chan CW, Yorke J, Farrell C, Bandla A, Ang E, Lopez V, Sundar R, Chan A. Minimal clinically important difference of the EORTC QLQ-CIPN20 for worsening peripheral neuropathy in patients receiving neurotoxic chemotherapy. Support Care Cancer. 2019 Dec;27(12):4753-4762. doi: 10.1007/s00520-019-04771-8. Epub 2019 Apr 10. PMID 30972646
- [Background] Molassiotis A, Cheng HL, Lopez V, Au JSK, Chan A, Bandla A, Leung KT, Li YC, Wong KH, Suen LKP, Chan CW, Yorke J, Farrell C, Sundar R. Are we mis-estimating chemotherapy-induced peripheral neuropathy? Analysis of assessment methodologies from a prospective, multinational, longitudinal cohort study of patients receiving neurotoxic chemotherapy. BMC Cancer. 2019 Feb 8;19(1):132. doi: 10.1186/s12885-019-5302-4. PMID 30736741
- [Background] Le-Rademacher J, Kanwar R, Seisler D, Pachman DR, Qin R, Abyzov A, Ruddy KJ, Banck MS, Lavoie Smith EM, Dorsey SG, Aaronson NK, Sloan J, Loprinzi CL, Beutler AS. Patient-reported (EORTC QLQ-CIPN20) versus physician-reported (CTCAE) quantification of oxaliplatin- and paclitaxel/carboplatin-induced peripheral neuropathy in NCCTG/Alliance clinical trials. Support Care Cancer. 2017 Nov;25(11):3537-3544. doi: 10.1007/s00520-017-3780-y. Epub 2017 Jun 20. PMID 28634656